CLINICAL TRIAL: NCT00288938
Title: Dermoscopic Diagnosis, Histopathological Correlation, and Cellular Immortalization of Melanocytic Nevi and Primary Cutaneous Melanoma
Brief Title: Natural History Study of Moles and Suspicious Melanoma
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060060; 06-C-0060; NCT00335530 (obsolete NCT alias)
Record Dates: First submitted 2006-02-08; First posted 2006-02-08 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-10-31

CONDITIONS: Melanocytic Nevi; Acquired Melanocytic Nevi; Primary Cutaneous Melanoma
Keywords: Suspicious mole; Congenital Nevus; Skin Cancer; Moles; Pigmented lesion; LCMN
MeSH Terms: conditions — Nevus, Pigmented; Skin Neoplasms; Nevus

SUMMARY:
Background:

* Melanocytic nevi, or "moles," are non-cancerous growths of a type of skin cell called a melanocyte.
* Large congenital melanocytic nevi (LCMN) are a special type of mole that begins to grow before birth and is larger than moles that develop after birth.
* Determining how melanocytes in moles and LCMNs differ from normal melanocytes may increase the ability to predict whether a mole will give rise to a melanoma (a type of skin cancer)

Objectives:

* To understand how melanomas develop, by studying moles, LCMNs, and pigmented skin lesions that are suspicious for melanoma
* To develop better criteria for diagnosing melanoma, particularly by using a device called a digital dermatoscope (a special camera, connected to a computer, that takes pictures of moles when they are magnified and illuminated)

Eligibility:

* Children 5 years old or older with an LCMN
* Adults 18 years old or older with 100 or more moles larger than 2 mm in diameter and at least one 4 mm or more
* Adults 18 years old or older with a pigmented lesion suspicious for melanoma

Design:

* Patients' personal and family health history is obtained.
* Patients are examined by investigative team doctors, and several lesions are examined with a dermatoscope.
* Additional photographs of part or all of the skin surface may be taken.
* Some lesions may be biopsied.
* Additional tests or examinations may be recommended.
* Patients are followed periodically for skin or physical examinations, photography, laboratory and imaging evaluations, and possible skin biopsies.
* Children may undergo brain magnetic resonance imaging (MRI)

DETAILED DESCRIPTION:
The objective of this study is to understand early transformation and malignant progression events of cutaneous melanoma by obtaining detailed clinical information and lesional tissue for analysis, cell culture, and immortalization from patients with melanocytic nevi, which frequently are precursor lesions of melanoma, and primary melanoma. An important goal of this study is the acquisition of melanocytes from lager congential melanocytic nevi (LCMN) and acquired melanocytic nevi (AMN) for analysis, culture and experimental manipulation. We do not propose to acquire melanocytes from pigmented lesions suspected to represent primary melanoma because of the importance of preserving all lesional tissue required to render accurate histopathological diagnosis. However, another aim of the study is the development of enhanced clinical criteria for the diagnosis of primary cutaneous melanoma, particularly using digital epiluminescent skin microscopy, or dermoscopy, for pigmented lesion image acquisition and analysis. The close comparison of dermoscopic images of pigmented skin lesions suspicious for melanoma with lesional histopathology should be useful for expanding the knowledge base about how dermoscopy , a relatively new technique used to evaluate pigmented skin lesions, can be used to diagnose a pigmented skin lesion as benign or malignant. These detailed comparisons may also provide information about how specific visual features within the dermoscopic image field correlate with histologic features of the lesion. This information may be useful for future possible studies designed to predict accurately which portions of a primary malignant melanoma can be removed for esperimental study while retaining sufficient lesional information to guide further treatment and render an accurate prognosis.

The study population will consist of three categories of patients: (1) infants and children with large congenital melanocytic nevi, (2) adults with numerous (less than 100) melanocytic nevi, and (3) patients with primary malignant melanoma. Establishment of the Pigmented Lesion Clinic required for the execution of this protocol will provide a mechanism for the evaluation of patients with numerous or unusual pigmented lesions, and for the entry of eligible patients into ongoing therapeutic trials for malignant melanoma. As the study progresses, it is anticipated that a substantial amount of formalin-fixed nevus and primary melanoma tissue with a high-degree of clinical annotation will be collected. As a secondary objective , the availability of this collection will be useful to support studies designed to evaluate new markers and techniques for the diagnosis of melanoma and atypical nevi, and for incorporation into a tissue microarray that will be available to the melanoma research community for target foundation validation.

Background:

The molecular events resulting in melanocyte transformation and the development of early melanoma are incompletely understood. Risk factors for the development of melanoma include genetic, phenotypic and environmental risk factors and can overlap. Also, persons with large numbers of nevi face a higher risk of melanoma. These risk associations, combined with knowledge obtained from basic studies on the survival, differentiation, and proliferation of the melanocyte, can provide hints about the molecular mechanisms that underlie the development of nevi and melanoma.

In this study we plan to acquire lesional tissue from pigmented lesions and develop enhanced clinical criteria for the diagnosis of primary cutaneous melanoma, particularly using digital epiluminescent skin microscopy, or dermoscopy, for pigmented lesion image acquisition and analysis. This information may be useful for future possible studies designed to predict accurately which portions of a primary malignant melanoma can be removed for experimental study while retaining sufficient lesional information to guide further treatment and render an accurate prognosis.

Objectives:

To obtain tissue from benign melanocytic nevi and from large congenital melanocytic nevi (LCMN) for experimental study.

To refine culture and immortalization methods for melanocytes derived from melanocytic nevi, permitting in vitro expansion of these cells for functional study.

To correlate clinical and dermoscopic observations of primary melanomas with histopathology to establish standards for sampling primary melanomas in a possible future study.

Eligibility:

Infants/Children less than 5 years of age with large congenital melanocytic nevus (LCMN, diagnosed clinically or by biopsy) that is greater than 20 cm in any one dimension or that is greater than 8 cm in any one dimension involving the scalp.

Adults greater than 18 years of age with greater than 100 melanocytic nevi greater than 2 mm in diameter with at least one melanocytic nevus greater than 4 mm in longest dimension or with a current pigmented lesion clinically suspicious for primary melanoma.

Design:

This is a natural history protocol designed to enroll 110 subjects who will be evaluated and followed over the course of their disease.

ELIGIBILITY:
* INCLUSION CRITERIA:

Infants/Children

Must be less than or equal to 5 years.

Must have large congenital melanocytic nevus (LCMN, diagnosed clinically or by biopsy) that is greater than 20 cm in any one dimension or that is greater than 8 cm in any one dimension involving the scalp.

Must have outside referring physician.

OR

Adults

Must be greater than 18 years.

Must have greater than or equal to 100 melanocytic nevi greater than 2 mm in diameter.

Must have at least one melanocytic nevus greater than or equal to 4 mm in longest dimension.

Can have prior history of cutaneous or ocular malignant melanoma.

Must have outside primary physician.

OR

Adults

Must be greater than 18 years.

Must have a current pigmented lesion clinically suspicious for primary melanoma.

Must have outside primary physician.

AND

All patients, or in the case of infants and children their parents or legal guardians, must be able to understand and sign an informed consent.

EXCLUSION CRITERIA:

The patient does not meet the inclusion criteria.

Diagnosis of genetic syndrome associated with multiple lentigines or nevi (Peutz-Jeghers syndrome, Carney complex, turner syndrome, Noonan's syndrome).

Two or more first-degree relatives with history of cutaneous melanoma and familial atypical mole-melanoma syndrome phenotype.

Diagnosis of cancer-associated syndrome (xeroderma pigmentosum, type I neurofibromatosis, Li-Fraumeni syndrome).

Inability to tolerate surgical procedure due to bleeding diathesis or disorder or other cause as determined by principal investigator.

Patient is unwilling to consider elective biopsy of a melanocytic nevus.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-02-03; Study Completion 2011-10-31

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Bastian BC, Kashani-Sabet M, Hamm H, Godfrey T, Moore DH 2nd, Brocker EB, LeBoit PE, Pinkel D. Gene amplifications characterize acral melanoma and permit the detection of occult tumor cells in the surrounding skin. Cancer Res. 2000 Apr 1;60(7):1968-73. PMID 10766187
- [Background] Bastian BC, LeBoit PE, Hamm H, Brocker EB, Pinkel D. Chromosomal gains and losses in primary cutaneous melanomas detected by comparative genomic hybridization. Cancer Res. 1998 May 15;58(10):2170-5. PMID 9605762
- [Background] Bataille V, Grulich A, Sasieni P, Swerdlow A, Newton Bishop J, McCarthy W, Hersey P, Cuzick J. The association between naevi and melanoma in populations with different levels of sun exposure: a joint case-control study of melanoma in the UK and Australia. Br J Cancer. 1998;77(3):505-10. doi: 10.1038/bjc.1998.81. PMID 9472652